CLINICAL TRIAL: NCT06356376
Title: The Effects of Pain and Pain Relief on Peripheral Nerve Excitability
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: UAarhus_AGK_MNG_2
Record Dates: First submitted 2023-12-17; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-12

CONDITIONS: Analgesia
Keywords: Pain; Excitability; Microneurography; Autonomic nervous system
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Participants
  Interventions: Device: Heat Stimulation

INTERVENTIONS:
Device: Heat Stimulation — Heat stimulation at a painful, but to the subject tolerable level.

SUMMARY:
This study will assess changes in nerve excitability of C-fibers, and changes in sympathetic or parasympathetic tone, when the subject experiences pain and pain relief.

The investigators will continuously measure blood pressure, heart rate, respiration rate, gastric motility, sympathetic skin response and C-fiber excitability while using thermal stimuli before and after an analgesic.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Participants able to give informed consent.

Exclusion Criteria:

* Chronic pain conditions
* Neurological or Psychiatric disease
* Other major diseases
* Pain medication within the last 24 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Subjects
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
C-fiber excitability | Through study completion, an average of 6 months
  Changes in C-fiber excitability measured in latency changes after electrical stimulation with a paired pulse protocol compared to an unpaired electrical stimulus.

SECONDARY OUTCOMES:
Action potential duration (ms) | Through study completion, an average of 6 months
  Averaged analysis from repeated measures of a single nerve fiber signal.
Action potential amplitude (V) | Through study completion, an average of 6 months
  Averaged analysis from repeated measures of a single nerve fiber signal.
Heart-rate variability (ms) | Through study completion, an average of 6 months
  Comparison of heart-rate variability during experimental pain stimulation and during pain relief.
Blood pressure variability (mmHg) | Through study completion, an average of 6 months
  Changes in continuous blood pressure measurement averages during experimental pain stimulation and during pain relief..
Sympathetic Skin Response (V) | Through study completion, an average of 6 months
  Amplitude of Sympathetic skin response during pain stimulation and relief respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Pain Research Center, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No